CLINICAL TRIAL: NCT05401344
Title: The Objective Assessment and Characteristics of Dry Nose From Clinical Perspective
Status: Completed | Type: Observational
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: V 1.0
Record Dates: First submitted 2022-05-26; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2018-12

CONDITIONS: Diagnostic Self Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dry nose patients
  Interventions: Diagnostic Test: test strips,sponges and cold dry air test
- normal controls
  Interventions: Diagnostic Test: test strips,sponges and cold dry air test

INTERVENTIONS:
Diagnostic Test: test strips,sponges and cold dry air test — Test strips were used to evaluated the degree of dry nose, sponges were used to obtain the nasal secretion and cold dry air test was used to making diagnosis of vasomotor rihinitis.

SUMMARY:
In the present study, we propose objective diagnostic criteria for dry nose (DN) and investigate its characteristics. Questionnaires were completed by each participant during recruitment to record demographic data. DN test strips were used to evaluate the severity of DN at five time points and allergic status was assessed based on serum sIgE levels. Nasal secretions were collected and vasomotor rhinitis was diagnosed using the cold dry air test. The diagnosis of allergic rhinitis (AR) was based on the criteria of the Allergic Rhinitis and its Impact on Asthma consensus statement. Data are expressed as median and interquartile range, unless otherwise specified. Statistical significance was set at P < 0.05. The reference range (RR) of the 5th, 10th, 25th, 50th, 75th, 90th, and 95th percentiles were determined for each test strip length at each time point. This study aimed to investigate the characteristics of and propose objective diagnostic criteria for DN.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of dry nose patients.

Exclusion Criteria:

* chronic rhinosinusitis and/or nasal polyposis, allergic fungal rhinosinusitis, immunological disease, tumor patients, pregnant women.

Ages: 23 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Overall, 20 patients (13 men and seven women) with dry nose and 100 controls (47 men and 53 women) were recruited for the study. The ages of the participants ranged from 23 to 73 years (mean = 47.7 years).
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2021-07-24 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
The length of the test strip. | 5 minutes
  We propose that the diagnostic criterion for DN is a strip length less than 17.0 mm at 5 min.

CONTACTS AND LOCATIONS:
Locations (1):
- Yifan Meng, Beijing, Beijing Municipality, China